CLINICAL TRIAL: NCT02080780
Title: Phase 1, Open-label, Drug-drug Interaction Study to Evaluate the Interaction Potential of Clarithromycin XL on Diltiazem Hydrochloride Cream 2% in Healthy Subjects
Brief Title: Study to Evaluate the Interaction Potential of Clarithromycin XL on Diltiazem Hydrochloride Cream 2% in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ventrus Biosciences, Inc (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN307-DDI-001
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: CLARITHROMYCIN/DILTIAZEM [VA Drug Interaction]
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2% Diltiazem & Clarithromycin XL (Experimental): 3 parts:
  1. - Single Dose, Diltiazem (Day 1)
  2. - Multiple Dose, Clarithromycin XL (Days 4-9)
  3. - Single Dose, Diltiazem (Day 8)
  Interventions: Drug: Clarithromycin XL; Drug: 2% Diltiazem

INTERVENTIONS:
Drug: Clarithromycin XL — Clarithromycin XL administered once daily on Days 4 through 9 as 2 x 500 mg tablets, 1000 mg per day, for a total of 6000 mg
Drug: 2% Diltiazem — 2% Diltiazem Hydrochloride Cream applied on Day 1 & Day 8 to the perianal area (~2.5 cm [1 inch]; ~8.5 mg)

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction potential of clarithromycin XL on Diltiazem hydrochloride (DTZ) 2% cream.

DETAILED DESCRIPTION:
This study was designed to investigate the potential effect of clarithromycin XL at steady state (administered orally, once daily on Days 4 through 9 as 2 x 500 mg tablets, 1000 mg per day, for a total of 6000 mg) on the PK of a single topical dose of diltiazem hydrochloride 2% cream applied to the perianal area (~2.5 cm [1 inch]; ~8.5 mg). This was a Phase 1 study with a single treatment arm. Efficacy was not assessed; therefore the study was of open-label design.

ELIGIBILITY:
Inclusion Criteria:

1. Were healthy subjects (as confirmed by medical history, laboratory work, and physical exam);
2. Were between 18 and 60 years of age, inclusive;
3. If of childbearing potential, were using an acceptable form of birth control (ie, nonhormonal intra-uterine device, diaphragm, condom, bilateral tubal ligation, abstinence, or were in a monogamous relationship with a partner who had a vasectomy);
4. In the case of females of childbearing potential, had a negative serum pregnancy test (SPT) at Screening and a negative urine pregnancy test (UPT) at Study Day -1, (a woman was considered to be of childbearing potential unless she was postmenopausal for at least 12 months or was surgically sterile [hysterectomy, bilateral oophorectomy]);
5. Had clinical lab tests (hematology, chemistry, and urinalysis), an electrocardiogram (ECG), and vital signs within normal limits, or assessed by the investigator as not of clinical significance; and
6. Were able to read, understand, and provide signed informed consent.

Exclusion Criteria:

1. On any drug treatment at the time of the study;
2. Had donated plasma (500 mL) within 7 days prior to drug administration;
3. Had donated or lost whole blood (excluding the volume of blood that was to be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration;
4. Were using and were unwilling to stop any other concomitant topical preparations in or around the anus and perianal area from Day -1 through the end of the study;
5. Had a hypersensitivity or allergy to the investigational compound/compound class used in this study, and bacterial fighting medications, including but not limited to clarithromycin XL , azithromycin, telithromycin, and erythromycin or to calcium channel blockers;
6. Had a history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease, that, in the opinion of the investigator, could have interfered with the study conduct or observation;
7. Were unable to adhere to or understand the requirements of the protocol;
8. Had a body mass index > 40 kg/m2;
9. Had a screening ECG >470 QTCF for females and >450 QTCF for males;
10. Were on active treatment with anti-viral therapies (eg, indinavir, nelfinavir, ritonavir) for human immunodeficiency virus (HIV);
11. Had been treated with any of the following medications within 14 days prior to signing the ICF:

    * CYP450 inhibitors and inducers;
    * CYP3A4 substrates, inhibitors, and inducers;
    * Benzodiazepines;
    * β-adrenoceptor antagonists (beta-blockers);
    * Calcium channel blockers;
    * Digoxin;
    * Investigational agents;
    * Opioids.
12. Had any of the following concomitant disease states:

    * Sick sinus syndrome except in the presence of a functioning ventricular pacemaker;
    * Second-or third-degree atrioventricular block except in the presence of a functioning ventricular pacemaker;
    * Hypotension (< 90 mm Hg systolic);
    * Acute myocardial infarction and pulmonary congestion documented by x-ray;
    * History of clinically significant renal disease;
    * History of clinically significant Alzheimer's or Parkinson's disease;
    * History of clinically significant hepatic disease;
    * Current infection treated with a macrolide antibiotic;
    * Clinical evidence or history of fecal incontinence;
    * Clinical evidence or history of anal fistula;
    * Clinical evidence or history of anal abscess;
    * History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis);
    * History of any prior anal or rectal surgery including but not limited to: lateral sphincterotomy and anal stretch;
13. Had a major organ transplant;
14. Had a serious illness in the 4 weeks preceding the beginning of treatment (ie, that resulted in missed work or hospitalization);
15. Had received treatment for any type of internal cancer within the 5 years prior to enrollment;
16. Had, in the opinion of the investigator, clinically significant abnormal clinical laboratory results at the time of screening;
17. Were females who were pregnant, were planning to become pregnant during the study, or were breastfeeding a child;
18. Were currently using narcotics chronically;
19. Were currently a smoker;
20. Had used an investigational drug or had participated in an investigational study within 30 days prior to dosing;
21. Had used prescription medication within 14 days prior to administration of study medication or over-the-counter (OTC) products (including natural food supplements vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption;
22. Were an employee, family member, or student of the investigator or clinical site;
23. Had any food allergy, intolerance, restriction, or special diet that, in the opinion of the investigator, could have contraindicated the subject's participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Paramus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% Diltiazem & Clarithromycin XL: 3 parts:
  1. - Diltiazem Single Dose
  2. - Clarithromycin XL (Days 4-9)
  3. - Diltiazem Single Dose after Clarithromycin
  Clarithromycin XL: Clarithromycin XL administered once daily on Days 4 through 9 as 2 x 500 mg tablets, 1000 mg per day, for a total of 6000 mg
  2% Diltiazem: 2% Diltiazem Hydrochloride Cream applied on Day 1 & Day 8 to the perianal area (~2.5 cm [1 inch]; ~8.5 mg)
Period: Overall Study
Arm/Group | 2% Diltiazem & Clarithromycin XL
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2% Diltiazem & Clarithromycin XL
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of 2% Diltiazem
Description: To evaluate the drug-drug interaction potential of clarithromycin XL on Diltiazem hydrochloride (DTZ) 2% cream.
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: ng / mL
Groups:
- Diltiazem Single Dose: On the morning of Day 1, subjects received a single dose of DTZ 2% cream (~2.5 cm [1 inch] strip of cream containing approximately 8.5 mg DTZ) applied perianally. area (~2.5 cm [1 inch]; ~8.5 mg)
- Diltiazem Single Dose After Clarithromycin: 2% Diltiazem Hydrochloride Cream applied on Day 8 to the perianal area (~2.5 cm [1 inch]; ~8.5 mg) following Clarithromycin XL administered once daily on Days 4 through 9 as 2 x 500 mg tablets, 1000 mg per day, for a total of 6000 mg
Arm/Group | Diltiazem Single Dose | Diltiazem Single Dose After Clarithromycin
Number analyzed (Participants) | 24 | 24
ng / mL | 0.340 (0.299) | 0.624 (0.475)

ADVERSE EVENTS:
Groups:
- Clarithromycin XL (Days 4-9): On Days 4 through 9, subjects received once daily doses of clarithromycin XL (2 tablets, 500 mg/tablet, total dose = 1000 mg/day; 6000 mg total in 6 days) with 24 hours between doses.
Arm/Group | Diltiazem Single Dose | Clarithromycin XL (Days 4-9) | Diltiazem Single Dose After Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 3/24 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diltiazem Single Dose (N=24) | Clarithromycin XL (Days 4-9) (N=24) | Diltiazem Single Dose After Clarithromycin (N=24)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less